CLINICAL TRIAL: NCT00621400
Title: A Multicenter Phase I/II Dose Escalation Study of Lenalidomide in Combination With Melphalan and Dexamethasone in Subjects With Newly-diagnosed Light-chain (AL)-Amyloidosis
Brief Title: Lenalidomide in Combination With Melphalan and Dexamethasone in Newly-diagnosed Light-chain (AL)-Amyloidosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Anne Omnes, Cellule Promotion Recherche Clinique
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD 07/7-G; EudraCT 2007-004739-43
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2010-05

CONDITIONS: Amyloidosis
Keywords: newly-diagnosed light-chain (AL)-amyloidosis
MeSH Terms: conditions — Amyloidosis; Immunoglobulin Light-chain Amyloidosis | interventions — Lenalidomide; Melphalan; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lenalidomide — 5 mg/day, orally for 21 days with 7 days rest (28 day cycle) for the first cohort; or 10mg/day, orally for 21 days with 7 days rest (28 day cycle) for the second cohort, 15mg/day, orally for 21 days with 7 days rest (28 day cycle) for the third cohort or 20mg/day, orally for 21 days with 7 days rest (28 day cycle) for the last and fourth cohort
  Other Names: Revlimid
Drug: Melphalan — 0,18mg/Kg/day from day 1- 4
  Other Names: Alkeran
Drug: Dexamethasone — 40mg/day from day 1- 4.

SUMMARY:
Amyloidosis results from tissue deposition of amyloid protein, composed mainly by the fragments of monoclonal immunoglobulin heavy chains or light chains. Accumulation of amyloid protein progressively disrupts normal tissue structure and ultimately leads to organ failure, most frequently in the kidneys, heart, liver and peripheral nervous system. A recently completed French prospective randomized trial, in patients presenting with newly AL-amyloidosis, compared two treatment regimens at the time of diagnosis: Melphalan-dexamethasone (conventional oral treatment), versus high dose of Melphalan followed by autologous stem cell transplantation (ASCT) (1). High-dose therapy was not associated with a better outcome. Melphalan-dex given monthly can be considered as the current standard of care, with a median survival of 56 months. The use of a combination of lenalidomide and dexamethasone has already been tested in patients with AL-amyloidosis (2). The initial dose of lenalidomide at 25 mg/day was poorly tolerated. However, a 15 mg/day dose regimen was well tolerated and effective, with an overall hematologic response rate of 67%. Hematologic responses were associated with clinical responses. Dispenzieri et al confirmed that the combination of Lenalidomide + dexamethasone achieved a 75% hematologic response rate, with a 42% organ response, and a median follow-up of 17 months in patients still receiving treatment (2006). These authors also recommended a lower dose of 15mg/day. The rationale for the present investigation is that addition of lenalidomide to the current standard of care (Melphalan-dexamethasone) might improve the hematologic response rate and the organ response rates both associated with a prolonged survival in patients with AL-amyloidosis. As the toxicity of the combination of M-dex + lenalidomide is unknown in patients with AL-amyloidosis, the dose of lenalidomide will start from the lowest one available, i.e., 5 mg/day and increased from 5 to 5 mg up to a maximum dose of 15 mg in combination with M-dex in 3 consecutive cohorts of patients, according to toxicity. When the optimal dose of lenalidomide will be defined, 9 additional patients will be included in the trial at the recommended dose-level to assess the feasibility of the combination M-dex-lenalidomide.

ELIGIBILITY:
Inclusion Criteria:

* De novo systemic biopsy proven AL-amyloidosis.
* Measurable organ site involvement consistent with the diagnosis.
* Adequate organ function defined as

  * Absolute neutrophil count > 1.0 x 109/L;
  * platelet count > 100x109/L;
  * AST (SGOT) and ALT (SGPT) < 2 x UNL;
  * Total bilirubin £ 1.5 mg/dL ;
  * creatinin serum level <150µmol/L (1.5mg/dl);
* Evaluable immunochemical abnormalities, including abnormal serum free light chain assay with an increase of either kappa or lambda light chain level.
* ECOG performance status of £ 2 at study entry (see Appendix BB).
* Age between18 and 70 years at the time of signing the informed consent form.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL at screening visit and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. See Appendix: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
* Able to understand and voluntarily sign an informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Able to take antithrombotic medicines such as low molecular weight heparin or warfarin (if needed).
* Disease free of prior malignancies for > 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* Subjects affiliated with an appropriate social security system.

Exclusion Criteria:

* Symptomatic multiple myeloma: multiple myeloma with related organ of tissue impairment (ROTI) according to the International Myeloma Working Group (16)
* Any other uncontrolled medical condition or comorbidity that might interfere with subject's participation.
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
* Use of any other experimental drug or therapy within 28 days of baseline.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Any prior treatment for amyloidosis.
* Known positive for HIV or infectious hepatitis, type A, B or C.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Determination of MTD by evaluation of hematological and non hematological toxicity
  The primary endpoint is to evaluate the incidence of dose limiting toxicities (DLT) during the first cycle of lenalidomide at a given dose level in order to determine the maximal tolerated dose (MTD) in a dose escalating study design.

SECONDARY OUTCOMES:
Complete (CR) or partial (PR) response, according to criteria defined during the 10th International Symposium on Amyloidosis
  To determine the hematologic response
disease progression from the date of the first dose to the date of the first observation of organ disease progression and observation of response
  To determine the rate of organ response
Value of frequent measurements of free light chain assays
  To determine interest of frequent measurments of free light chain assays for patients
Incidence of Treatment Emergent Adverse Event (TEAE), Serious Adverse Event (SAE) and laboratory abnormalities
  To assess the safety profile of the combination therapy
time between first documentation of hematologic response and disease progression
  To measure hematological duration
disease progression from the date of the first dose to the date of the first observation of hematologic disease progression
  Time to hematologic disease progression

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - CHRU d'Amiens, Amiens
  - CHRU de Lille, Lille
  - CHU de Limoges, Limoges
  - CHU de Nantes, Nantes
  - Hôpital Saint-Louis, Paris
  - Hôpital Pitié Salpetrière, Paris
  - Hôpital necker, Paris
  - Hôpitaux Civils de Lyon, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes
  - CHU de Toulouse, Toulouse
  - CHRU deTours, Tours

REFERENCES:
- [Derived] Moreau P, Jaccard A, Benboubker L, Royer B, Leleu X, Bridoux F, Salles G, Leblond V, Roussel M, Alakl M, Hermine O, Planche L, Harousseau JL, Fermand JP. Lenalidomide in combination with melphalan and dexamethasone in patients with newly diagnosed AL amyloidosis: a multicenter phase 1/2 dose-escalation study. Blood. 2010 Dec 2;116(23):4777-82. doi: 10.1182/blood-2010-07-294405. Epub 2010 Aug 19. PMID 20724537